CLINICAL TRIAL: NCT05000151
Title: Lung Volume Perception and Impact of a Cognitive Task on Ventilation in Healthy Subjects and Subjects With Hypermobile Ehlers-Danlos Syndrome.
Brief Title: Lung Volume Perception and Impact of a Cognitive Task on Ventilation in Hypermobile Ehlers-Danlos Syndrome.
Acronym: ProprioRespi
Status: Completed | Type: Observational
Sponsor: Hakimi Adrien (Other)
Responsible Party: Sponsor-Investigator, Hakimi Adrien, MCs, PT, Clinique de la Mitterie
Organization: Clinique de la Mitterie (Other)
Other Study IDs: ProprioRespi
Record Dates: First submitted 2021-07-30; First posted 2021-08-11 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hypermobile Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Hypermobile Ehlers-Danlos patients (n=21)
- Healthy subjects: Healthy subjects recruited from the clinic's staff (n=21) Age, Gender and BMI matched with hEDS patients

SUMMARY:
Patients with hypermobile Ehlers-Danlos syndrome have respiratory and proprioceptive disorders. The aim of this study is to explore whether there is an alteration in lung volume perception in patients with hEDS compared to healthy subjects, and whether a cognitive task can influence ventilation control differently in subjects with hEDS than in healthy subjects.

ELIGIBILITY:
Inclusion Criteria (common):

* More than 18 years old
* Understanding French

Inclusion Criteria (hEDS Patients):

* hEDS diagnosis

Inclusion Criteria (healthy subjects):

* Age (±5 years), Gender and BMI (±2.5kg/m²) matching

Exclusion Criteria (common):

* Pregnancy

Exclusion Criteria (hEDS Patients):

* Respiratory comorbidity independent of hEDS
* Previous participation in a rehabilitation programme at the clinic

Exclusion Criteria (healthy subjects):

* Known respiratory or proprioceptive pathology
* Hypermobility (evaluated with the Beighton score)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited through practitioners working with the clinic, who will propose participation in the study during consultations with patients diagnosed with EDS.
  The recruitment of subjects for the control group will be carried out by internal communication within the Clinique de la Mitterie on a voluntary basis.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Accuracy of lung volume perception | Baseline
  The perception of lung volume is assessed using a device comprising a flow meter, an electronic acquisition card and an LCD screen. Subjects will be given 3 trials to train to perceive a target lung volume and then 3 trials without feedback to reproduce that target lung volume. The mean of the absolute deviations from the target volumes in percent is used as the primary outcome.

SECONDARY OUTCOMES:
Minute ventilation with or without cognitive task | Baseline
  The minute ventilation will be calculated over 1 minute without cognitive task and then over 1 minute with cognitive task (trail making test part B).
Respiratory rate variability | Baseline
  The time interval between each inspiratory peak will be recorded and will allow the calculation of the standard deviation and the root mean square with and without the cognitive task.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille Bergoin, MD, Principal Investigator — Clinique de la Mitterie; Patrick Mucci, Prof., Study Director — UREPSSS
Locations (1):
- Clinique de la Mitterie, Lomme, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hakimi A, Bergoin C, De Jesus A, Hermand E, Fabre C, Mucci P. Impairment of lung volume perception and breathing control in hypermobile Ehlers-Danlos syndrome. Sci Rep. 2024 Apr 6;14(1):8119. doi: 10.1038/s41598-024-58890-2. PMID 38582758